CLINICAL TRIAL: NCT02706730
Title: A 6-Month, Multicenter, Phase 3, Open-Label Extension Safety Study of OTO-104 Given At 3-Month Intervals by Intratympanic Injection in Subjects With Unilateral Meniere's Disease
Brief Title: A 6-Month Extension Study of OTO-104 in Meniere's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Negative Efficacy Results from the recently completed Phase 3 study 104-201506
Sponsor: Otonomy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104-201509
Record Dates: First submitted 2016-03-08; First posted 2016-03-11 (Estimated); Results first posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-11

CONDITIONS: Meniere's Disease
MeSH Terms: conditions — Meniere Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OTO-104 (Experimental): 12 mg dexamethasone
  Interventions: Drug: OTO-104

INTERVENTIONS:
Drug: OTO-104 — Single intratympanic injection of 12 mg OTO-104

SUMMARY:
This is an open-label extension study of a single intratympanic injection of OTO-104 given every 3 months for a total of 2 injections. Subjects must have completed either Otonomy study 104-201102 (Phase 2b study of OTO-104) or 104-201506 (Phase 3 study of OTO-104) in order to be eligible for this open-label extension study.

ELIGIBILITY:
Inclusion Criteria includes, but is not limited to:

* Subject has completed the OTO-104 Phase 2b (104-201102) or Phase 3 (104-201506) clinical study.
* Subject has a diagnosis of definite unilateral Meniere's disease by 1995 AAO-HNS criteria

Exclusion Criteria includes, but is not limited to:

* Subject is pregnant or lactating.
* Subject has a history of immunodeficiency disease.
* Subject has experienced an adverse reaction to intratympanic injection of steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathie Bishop, PhD, Study Chair — Otonomy, Inc.
Locations (1):
- Many sites in US. Refer to the contact info listed below., San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 189 subjects registered for this study and signed informed consent and were enrolled. Of the 189 subjects enrolled, 49 had previously completed the 104-201102 study and 140 had previously completed the 104 201506 study. The first subject enrolled on February 16, 2016, and the last subject completed on September 9, 2017.
Pre-assignment Details: This study was terminated early based on results of study 104-201506, a US Phase 3 study that indicated no statistically significant difference in the primary endpoint of reduction in definitive vertigo days (DVD) for OTO-104 vs placebo nor for any of the secondary endpoints. Decision was made to terminate all ongoing studies on August 31, 2017, including this study. At the time of termination, 156 subjects completed the study through Month 3 and 121 subjects completed the study through Month 6.
Groups:
- OTO-104: Intratympanic injection of 12 mg OTO-104
Period: Overall Study
Arm/Group | OTO-104
Started | 189
Completed | 156
Not Completed | 33
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 5
Not completed — Withdrawal by Subject | 11
Not completed — Study Terminated by Sponsor | 11
Not completed — Subject chose not to receive injection | 3

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all subjects who received at least 1 dose of study drug.
Arm/Group | OTO-104
Number analyzed (Participants) | 189
Age, Continuous [Median (Full Range); unit: years] | 57.0 [24 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 176
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 179
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 189
Duration of Meniere's disease [Count of Participants; unit: Participants]
  ≤5 years | 125
  6-10 years | 28
  11-15 years | 22
  >15 years | 14

OUTCOME MEASURES:

1. Primary Outcome: Otoscopic Examination - Tympanic Membrane Perforation at Week 24 (Month 6)
Description: Otoscopic examinations were conducted at each visit. It was considered important to understand if the tympanic perforation that resulted from the IT injection persisted at the end of study visit (Week 24 [Month 6]).
Time Frame: 6 Months
Population: The 6-month Safety Analysis Set included all subjects who received at least 1 dose of study drug and completed the study at the Month 6 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | OTO-104
Number analyzed (Participants) | 121
Participants
  Perforation present: pinhole size | 4
  Perforation present: ≤25% tympanic membrane | 3
  Perforation present: ≤25% tympanic membrane Perforation present: >25% and ≤50% tympanic membrane | 1
  Perforation present: %50 tympanic membrane | 0
  Not Present | 113

ADVERSE EVENTS:
Time Frame: Reported or observed during or after dosing with the study drug up until end of study (Month 6).
Arm/Group | OTO-104
All-Cause Mortality (participants affected / at risk) | 1/189
Serious Adverse Events (participants affected / at risk) | 7/189
Other Adverse Events (participants affected / at risk) | 30/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTO-104 (N=189)
Hemiplegic Migraine (Nervous system disorders) | 1 (1)
Omental Infarction and Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Acute Myeloid Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Angina Pectoris (Cardiac disorders) | 1 (1)
Deafness, Unilateral (Ear and labyrinth disorders) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTO-104 (N=189)
Vertigo (Ear and labyrinth disorders) | 7 (7)
Tinnitus (Ear and labyrinth disorders) | 6 (6)
Ear Pain (Ear and labyrinth disorders) | 4 (4)
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 4 (4)
Dizziness (Nervous system disorders) | 5 (5)
Suicidal Ideation (Psychiatric disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT02706730/Prot_SAP_000.pdf